CLINICAL TRIAL: NCT05247528
Title: A Phase 1B, Multiple Ascending Dose Trial Examining The Safety And Tolerability Of Subcutaneous MANP In Difficult To Control/Resistant Hypertensive Subjects
Brief Title: Safety And Tolerability Of Subcutaneous MANP In Difficult To Control/Resistant Hypertensive Subjects
Acronym: DTC/RHS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: E-Star BioTech, LLC (Industry)
Collaborators: Mayo Clinic (Other); Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ES_MANP_21-01
Record Dates: First submitted 2021-12-22; First posted 2022-02-21 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Resistant Hypertension; Difficult to Control Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator (Placebo Comparator): * Subjects randomized to the placebo arm, will receive a single subcutaneous injection each morning daily.
  * Intervention: Placebo
  Interventions: Drug: Placebo
- MANP (Experimental): * Subjects randomized to the experimental arm, will receive a single subcutaneous injection each morning daily. (multiple ascending dose cohorts)
  * Intervention: Drug: MANP
  Interventions: Drug: MANP

INTERVENTIONS:
Drug: MANP — Novel designer peptide to represent a pGC-A/cGMP therapeutic
  Arms: MANP
Drug: Placebo — Placebo Comparator
  Arms: Placebo Comparator

SUMMARY:
A randomized, double-blind, placebo-controlled multiple ascending dose study in hypertensive subjects on stable doses of at least three hypertensive drugs for at least 6 weeks prior to Screening. The study will consist of screening, PK-unit admittance, and safety follow up periods.

Subjects will be randomized at a 6:2 ratio of either MANP or placebo and will be stratified by race in each dosage cohort. The entire first Cohort will be given the lowest dosage with subsequent cohorts progressing sequentially to the higher doses depending on safety and tolerability of the previous cohort.

Endpoints not related to the safety reviews will be analyzed after the last patient last visit (LPLV).

ELIGIBILITY:
Inclusion Criteria:

* DTC/RH diagnosed with clinic SBP ≥140 mmHg or DBP ≥ 90 mmHg (or SBP ≥ 130 mmHg or DBP ≥ 80 mmHg for diabetics) while on at least three standard-of-care antihypertensive medications (which must include a diuretic).
* MDRD eGFR ≥ 30 mL/min.
* Men and women between the ages of 18 - 80.
* BMI within the range of 18-40 kg/m2.
* Women of childbearing potential must not be pregnant and agree to avoid becoming pregnant while receiving study treatment and for 14 days after the last study visit.

Exclusion Criteria:

* HbA1c ≥ 8% at Screening.
* Use of other investigational drugs within 30 days of screening or foreseen use during the study.
* Inability to comply with study requirements as judged by the Investigator.
* Pregnant and/or breastfeeding.
* Any disease or condition (medical or surgical) which, in the opinion of the investigator, might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of study drug, or would place the subject at increased risk.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events | through study completion, an average of 2 months.
  Number and percent of participants with one or more Treatment Emergent Adverse Events (TEAEs) or any serious adverse events (SAEs).
Blood Pressure | From baseline to Days 1-6, Day 12, and 21.
  Change in SBP and DBP
Hematology Hematocrit | From baseline to Day 21.
  Change in Percent Hematocrit
Physical Examination: Body Parts | From baseline to Day 21
  Change in investigator assessment of the condition of body parts (head, throat, abdomen, and extremities)
ECG: QT interval | From baseline to Days 1-6 and Day 21.
  Change in 12-Lead ECG QT Interval
Temperature | From baseline to Days 1-6, Day 12, and 21.
  Change in Temperature
Pulse Rate | From baseline to Days 1-6, Day 12, and 21.
  Change in Pulse Rate
Hematology: Hemoglobin | From baseline to Day 21
  Change in g/dL Hemoglobin
Hematology: Mean Corpuscular Hemoglobin | From baseline to Day 21
  Change in the mean corpuscular hemoglobin.
Hematology: Platelets | From baseline to Day 21
  Change in platelet count
Hematology: RBC distribution | From baseline to Day 21
  Change in red blood cell distribution width
Hematology: RBC | From baseline to Day 21
  Change in red blood cell count
Hematology: WBC | From baseline to Day 21
  Change in white blood cell count
Chemistry: Sodium | From baseline to Day 21
  Change in Sodium concentration.
Chemistry: Potassium | From baseline to Day 21
  Change in Potassium concentration.
Chemistry: Chloride | From baseline to Day 21
  Change in Chloride concentration
Chemistry: Bicarbonate | From baseline to Day 21
  Change in Bicarbonate concentration
Chemistry: Alanine aminotransferase | From baseline to Day 21
  Change in ALT (IU/L)
Chemistry: Aspartate aminotransferase | From baseline to Day 21
  Change in AST (IU/L)
Chemistry: Alkaline phosphatase | From baseline to Day 21
  Change in Alkaline phosphatase (IU/L)
Chemistry: Bilirubin | From baseline to Day 21
  Change in Total bilirubin (mg/dL)
Chemistry: Blood urea nitrogen | From baseline to Day 21
  Change in BUN (mg/dL)
Chemistry: Creatinine | From baseline to Day 21
  Change in Creatinine (mg/dL)
Chemistry: Glucose | From baseline to Day 21
  Change in Glucose (mg/dL)
Chemistry: HbA1c | From baseline to Day 21
  Change in percent HbA1c
Physical Examination: Organs | From baseline to Day 21
  Change in investigator assessment of the condition of organs (skin, eyes, ears, nose, thyroid, lungs, liver, spleen, and lymph nodes)
Abbreviated Neurological Examination | From baseline to Day 21
  Change in investigator assessment of neurological condition
ECG: QTc interval | From baseline to Days 1-6 and Day 21
  Change in 12-Lead ECG QTc (Fridericia's) Interval

SECONDARY OUTCOMES:
Cardiac Metrics: Blood pressures | From Baseline for Day 1-6
  Change in SBP and DBP
Serum creatinine | From Baseline for Day 1-6
  Change in Serum creatinine
MANP | From baseline for Day 1 & Day 5
  Change in amount of Plasma MANP both in plasma.
Immune Response | From baseline for Day 1, Day 5, Day 12, & Day 21
  Change in amount of anti-MANP and anti-ANP
Metabolics | From baseline for Day 1 & Day 5
  Change in amount of non-esterified insulin and glucose.
eGFR, | From Baseline for Day 1-6
  Change in eGFR,
Urine flow rate | From Baseline for Day 1-6
  Change in urine flow rate
Urinary Sodium Excretion | From Baseline for Day 1-6
  Change in amount of urinary sodium excretion
cGMP | from baseline for Day 1 & Day 5
  Change in amount of cGMP both in plasma and urine
Aldosterone | from baseline for Day 1 & Day 5
  Change in amount of aldosterone both in plasma and urine
Cardiac Metrics: | From Baseline for Day 1-6
  Heart Rate

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Gonzalez, Study Director — E-Star
Locations (5):
- United States (5):
  - USA Clinical Site 03, Anniston, Alabama
  - USA Clinical Site 01, Tustin, California
  - USA Clinical Site 02, DeLand, Florida
  - USA Clinical Site 04, Decatur, Georgia
  - USA Clinical Site 05, Owensboro, Kentucky

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication